CLINICAL TRIAL: NCT01254721
Title: A Comparison of the Effectiveness of Seroquel XR and Seroquel XR Plus Lithium in Patients With Acute Bipolar Mania: An Open-label, Randomized, Parallel Groups, Rater-blinded, 4 Week, Multicenter, Comparative, Phase 4 Study
Brief Title: A Comparison of the Effectiveness of Seroquel XR and Seroquel XR Plus Lithium in Patients With Acute Bipolar Mania: An Open-label, Randomized, Parallel Groups, Rater-blinded, 4 Week, Multicenter, Comparative,Study
Acronym: STAR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty of recruitment.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00086
Record Dates: First submitted 2010-12-03; First posted 2010-12-07 (Estimated); Results first posted 2014-05-08 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Acute Bipolar Mania
Keywords: Acute bipolar mania; Seroquel XR; Seroquel XR plus lithium; Quetiapine fumarate
MeSH Terms: interventions — Quetiapine Fumarate; Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Seroquel XR tablet
  Interventions: Drug: Quetiapine fumarate
- 2 (Active Comparator): Seroquel XR + lithium
  Interventions: Drug: Quetiapine fumarate; Drug: lithium

INTERVENTIONS:
Drug: Quetiapine fumarate — eXtended Release(XR) 50mg, 200mg, 300mg and/or 400mg tablet, oral, once daily in the evening, from assignment to the end of the study.
Drug: lithium — 300mg tablet, oral
  Arms: 2

SUMMARY:
The primary objective of this study is to compare the efficacy of Seroquel XR monotherapy compared with Seroquel XR plus lithium in the treatment of acute bipolar mania by evaluation of the changes from baseline in Young Mania Ratings Scale (YMRS) total score to Day 29 using the last observation carried forward method.

DETAILED DESCRIPTION:
A comparison of the effectiveness of Seroquel XR and Seroquel XR plus lithium in patients with acute bipolar mania: An open-label, randomized, parallel groups, rater-blinded, 4 week, multicenter, comparative, phase 4 study.

ELIGIBILITY:
Inclusion Criteria:

* Female and/or male inpatients or outpatients, aged over 18 years and under 65 years
* Documented clinical diagnosis meeting the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) criteria
* YMRS total score =20 at enrollment and randomization (Day 1) Patients had a history of at least one manic episode that required hospitalization and/or treatment with a mood stabilizer or antipsychotic.
* Female patients must have a negative urine human chorionic gonadotropin (HCG) test at enrolment and must be using a reliable method of birth control, ie, barrier method, oral contraceptive, implant, dermal contraception, long-term injectable contraceptive

Exclusion Criteria:

* Pregnancy or lactation Meeting the criteria for any other (than bipolar disorder) DSM-IV Axis I diagnosis, concomitant organic mental disorder or mental retardation
* Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
* Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomization/baseline
* Known intolerance or hypersensitivity to, or lack of response to previous treatment with quetiapine fumarate or lithium

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2010-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yeon Ho Joo, Principal Investigator — Asan Medical Center, St. Asan medical center 86, Songpa-gu, Seoul Korea
Locations (5):
- South Korea (5):
  - Research Site, Ansan, Gyeonggi-do
  - Research Site, Daegu, Gyeongsangbuk-do
  - Research Site, Jinju, Gyeongsangnam-do
  - Research Site, Pusan, Gyeongsangnam-do
  - Research Site, Seoul, Seoul

RESULTS

PARTICIPANT FLOW:
Groups:
- Seroquel XR: Seroquel XR: 300mg, After that, 400mg to 800mg, Study medication will be administered orally, once daily in the evening.
  Treatment duration: 28 days
- Seroquel XR + Lithium: Seroquel XR: 300mg, After that, 400mg to 800mg Study medication will be administered orally, once daily in the evening Lithium will be started with 300mg tid on Day 1 then adjusted between the 900mg/day and 1200mg/day from Day 2 within lithium concentration [0.8~1.2mEq/L].
  Treatment duration: 28 days
Period: Overall Study
Arm/Group | Seroquel XR | Seroquel XR + Lithium
Started | 67 (Seroquel XR: 300mg) | 64 (Seroquel XR: 300mg Lithium: 900mg)
Completed | 52 | 42
Not Completed | 15 | 22
Not completed — Lost to Follow-up | 0 | 4
Not completed — Lack of Efficacy | 4 | 2
Not completed — Death | 0 | 1
Not completed — technical problum | 1 | 0
Not completed — Adverse Event | 2 | 3
Not completed — Withdrawal by Subject | 8 | 11
Not completed — Wrongly randomization | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Seroquel XR | Seroquel XR + Lithium | Total
Number analyzed (Participants) | 63 | 58 | 121
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age in ITT population.
  Years
    Age | 38.4 (9.8) | 36.9 (11.7) | 37.7 (10.7)
Age, Customized [Mean (Standard Deviation); unit: Years] — Age at onset of acute bipolar mania in ITT analysis set
  Years
    Age at onset of acute bipolar mania | 31.0 (10.6) | 30.0 (11.3) | 30.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Total ITT analysis set is 121
  Participants
    Female | 37 | 34 | 71
    Male | 26 | 24 | 50
Total No. of acute bipolar mania episodes over lifetime [Mean (Standard Deviation); unit: Episodes] | 4.24 (4.31) | 3.25 (2.42) | 3.76 (3.54)
Bipolar I Disorder [Number; unit: Number of Patients in ITT analysis set] — number of patients experiencing manic and mixed episodes in ITT analysis set
  Number of Patients in ITT analysis set
    Manic Episodes | 57 | 51 | 108
    Mixed Episodes | 6 | 7 | 13

OUTCOME MEASURES:

1. Secondary Outcome: The Change From Baseline up to Day 29 and Final Assessment in the Clinical Global Impression-Severity of Illness Scale (CGI-S)
Description: The Severity of Illness scale (CGI-S) is scored to rate the patient's current clinical state. The score range is form 0 to 7. A CGI-S score of 1 indicates that a patient is "Normal, not at all ill" and a score of 7 indicates that a patient is "Among the most extremely ill patients".
Time Frame: From Baseline to Day 29
Measure: Mean (Standard Deviation); unit: scores on the scale
Arm/Group | Seroquel XR | Seroquel XR + Lithium
Number analyzed (Participants) | 63 | 58
scores on the scale | -1.37 (1.52) | -1.58 (1.56)

2. Primary Outcome: The Changes From Baseline in Young Mania Rating Scale (YMRS) Total Score to Day 29
Description: The Young Mania Rating Scale (YMRS) is an eleven-item, multiple-choice diagnostic questionnaire which psychiatrists use to measure the severity of manic episodes. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. These four items are given twice the weight of the others to compensate for poor cooperation from severely ill patients. Total score is summed of 11items. Total score rage is from 0 to 60 and the higher score represent a worse oucome.
Time Frame: From Baseline to Day 29
Measure: Mean (Standard Deviation); unit: scores on the scale
Arm/Group | Seroquel XR | Seroquel XR + Lithium
Number analyzed (Participants) | 63 | 58
scores on the scale | -13.7 (13.8) | -15.5 (13.3)

ADVERSE EVENTS:
Time Frame: Day1 to Day29
Description: Safety set number is 130 (Seroquel XR 68 and Seroquel XR+Lithium 62)
Arm/Group | Seroquel XR | Seroquel XR + Lithium
Serious Adverse Events (participants affected / at risk) | 2/68 | 2/62
Other Adverse Events (participants affected / at risk) | 52/68 | 49/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Seroquel XR (N=68) | Seroquel XR + Lithium (N=62)
MANIC SYMPTOMS AGGRAVATION (Psychiatric disorders) | 0 (0) | 1 (1)
BIPOLAR MANIA (Psychiatric disorders) | 1 (1) | 0 (0)
MOOD ELEVATION (Psychiatric disorders) | 1 (1) | 0 (0)
DEATH (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Seroquel XR (N=68) | Seroquel XR + Lithium (N=62)
Headache (Nervous system disorders) | 6 (6) | 6 (10)
Dyspepsia (Gastrointestinal disorders) | 8 (9) | 3 (4)
Dry mouth (Gastrointestinal disorders) | 3 (4) | 7 (7)
Nasopharyngitis (Infections and infestations) | 5 (6) | 5 (5)
Insomnia (Psychiatric disorders) | 8 (8) | 2 (2)
Constipation (Gastrointestinal disorders) | 20 (21) | 20 (21)
Akathisia (Nervous system disorders) | 4 (4) | 5 (5)
Tremor (Nervous system disorders) | 3 (3) | 6 (6)
Dizziness (Nervous system disorders) | 6 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less